CLINICAL TRIAL: NCT05919602
Title: Effectiveness of Image Visualization in Reducing Preoperative Anxiety. Pilot Study
Brief Title: Effectiveness of Images in Reducing Preoperative Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: María del Mar Perez Saavedra (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor-Investigator, María del Mar Perez Saavedra, Principal investigator, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Organization: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EIRPA
Record Dates: First submitted 2023-03-07; First posted 2023-06-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Upper Limb Injury
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Subjects on the waiting list for upper limb surgery that on the day of surgery, only anxiety will be evaluated before the operation and no intervention would be performed before the operation.
- Intervention group (Experimental): Subjects on the waiting list for upper limb surgery on the day of surgery, anxiety will be evaluated before the operation and intervention would be performed before the operation.
  Interventions: Other: Visualization of an image catalogue

INTERVENTIONS:
Other: Visualization of an image catalogue — Participants in the intervention group will be shown a catalog consisting of 8 images, each for 8 seconds, 25 minutes before entering the operating room. The images shown will be landscapes and/or objects of nature as an expression of neutrality, with light and soft colors, and will be chosen by over 50% of the research team from a gallery of 20 possible images that meet the aforementioned requirements.
  Arms: Intervention group

SUMMARY:
Introduction: Current evidence supports the existence of preoperative anxiety and its undesirable effects during surgery and in the postoperative period. Despite numerous studies that have evaluated the effectiveness of different non-pharmacological interventions in reducing preoperative anxiety, we have not found any that use an image catalog.

Objective: To evaluate the effect of an intervention based on the visualization of an image catalog on the improvement of perceived anxiety in patients undergoing upper limb orthopedic surgery.

Methodology: A prospective, randomized, controlled, parallel-group clinical trial with a 1:1 ratio will be conducted. The study will include 167 patients scheduled for upper limb surgery who are over 18 years old, without blindness or decreased visual acuity that cannot be corrected with appropriate lenses. The subjects will be invited to explain the study's objective and perform baseline assessments. On the day of the surgical intervention, both groups will receive standard care, but those in the intervention group will also visualize a catalog of 8 images, 25 minutes before entering the operating room. In addition, 30 and 10 minutes before the intervention begins, all patients included in the study will have vital signs taken, be administered Spielberger's anxiety scale, visual analog scale for anxiety, and cortisol levels in saliva will be determined as measures of preoperative anxiety. The final evaluation will measure whether this intervention results in decreased anxiety, postoperative complications resulting from anxiety, and length of hospital stay.

DETAILED DESCRIPTION:
1. Design:

   This study will be a controlled and randomized clinical trial of two parallel groups aimed at evaluating the effect of showing a catalog of 8 images in reducing perceived anxiety in patients undergoing traumatic surgery of the upper limb.
2. Study setting:

   The study will be carried out in the specialized care area, specifically in the surgical block, in the Traumatology and Orthopedics Service of CAUSA (University Hospital Complex of Salamanca, Spain).
3. Study subjects:

Participants will be selected in Traumatology consultations by consecutive sampling among those who meet the selection criteria.

Inclusion criteria:

1. Individuals of both sexes over 18 years of age with upper limb pathology that will be surgically treated at CAUSA.
2. Signed informed consent.

Exclusion criteria:

1. Pathology to be surgically treated with a location other than the upper limb.
2. Patients with a score of less than 26 points on the Mini Mental Examination (MMSE).
3. Blind or visually impaired individuals who cannot correct their vision with appropriate lenses.
4. Any other circumstance at the discretion of the investigators.

4. Sample size: The final sample will consist of 167 subjects selected by simple random sampling from the patients treated in the Traumatology consultation at CAUSA who are going to undergo traumatic surgery of the upper limb.

These subjects will then be randomized in a ratio of 1:1 to control and intervention groups, using Epidat 4.2 software.

The sample size has been estimated taking into account the main variable of the study: reduction of preoperative anxiety according to the STAI scale, compared to standard care. Since no studies evaluating the reduction of preoperative anxiety using image visualization have been described, to calculate the sample size, we used the systematic review conducted by Bradt et al. (19), which obtained a reduction of 6 points on the aforementioned scale using another non-pharmacological method such as music therapy in reducing preoperative anxiety. Accepting a risk α of 0.05 and a risk β of 0.2, with a standard deviation of 2.2 points, 152 subjects (76 in each group) are needed to detect a decrease of at least 1 point in the STAI scale of the intervention group compared to the control group.

This estimate will be increased by 10% of subjects to cover possible losses throughout the study.

5. Study variables: Sociodemographic variables: Information on age, gender, marital status, educational level, with or without children, occupation, and employment status will be collected from all participants. Additionally, the existence of comorbidities and personal history, especially anxiety and depression, will be evaluated.

Clinical variables:

Blood pressure and heart rate: Blood pressure and heart rate will be measured in each participant during the baseline visit, as well as 30 and 10 minutes before surgery. An OMRON M10 IT® blood pressure monitor will be used, following current recommendations of the European Society of Hypertension.

Stress response marker: Cortisol quantification will be performed using the Elecsys Cortisol II Cobas® saliva test following the manufacturer's instructions (Roche). Three samples will be collected from each patient, specifically, one on the day of the baseline visit and the other two on the day of surgery, 30 and 10 minutes before entering the operating room.

Preoperative anxiety: This will be assessed using the Spanish validated version of the State-Trait Anxiety Inventory (STAI) scale by Spielberger. The scale used in the study distinguishes between anxiety as a state and anxiety as a personality trait. The scale consists of 40 items, 20 of which evaluate anxiety as a trait (A/T) and the other 20 evaluate anxiety as a state (A/S). State anxiety or momentary anxiety is characterized by subjectively perceived feelings of tension and apprehension, as well as by hyperactivity of the autonomic nervous system in response to a specific situation. In contrast, the characteristics of anxiety as a trait predispose the subject to perceive the world in a certain way and to manifest relatively stable response tendencies over time.

Participants are asked to respond to each item on a 3-point Likert scale. Then, the total value is calculated (possible range 0-60 for each questionnaire). The full 20 items that measure A/T and the 20 items that measure A/S will be administered during the baseline visit. On the day of surgery, only the scale related to A/S will be applied.

Additionally, anxiety will also be evaluated through the Visual Analog Anxiety Scale (VAAS) in adults, which consists of presenting a 100 mm line where the participant marks their level of anxiety at that moment, with the left end valued as "no anxiety" and the right end as "maximum anxiety". Similarly, it will be applied during the baseline visit and 30 and 10 minutes before entering the operating room on the day of surgery.

Procedure outcome variables: Complications derived from the procedure (pain and its control, infections, length of hospital stay, etc.) will be reviewed to evaluate whether the intervention reduces them.

6. Intervention performed:

Common intervention in both groups:

Participants will receive standard preoperative care.

Specific intervention in the experimental group:

Participants in the intervention group will be shown a catalog consisting of 8 images, each for 8 seconds, 25 minutes before entering the operating room. The images shown will be landscapes and/or objects of nature as an expression of neutrality, with light and soft colors, and will be chosen by over 50% of the research team from a gallery of 20 possible images that meet the aforementioned requirements.

7. Masking strategy: Due to the design of the study, the participant subjects and the person responsible for showing the catalog of images cannot be blinded. However, those responsible for analyzing the saliva samples and the statistician will be blinded.

8. Study procedure: Subjects who appear during the course of the study will be invited to participate during the interview conducted in the traumatology clinic. Subjects who are already on the waiting list for upper limb surgery will be invited to participate in the study by phone. Subsequently, the researchers will contact interested individuals, explain the purpose of the study, check inclusion and exclusion criteria, and arrange an interview.

At the baseline visit, the objective of the study, its procedures, risks, and expected benefits will be explained again, and the patient information sheet will be handed over along with the informed consent form. After signing the consent form, sociodemographic data, medical history, presence of comorbidities, and use of concomitant medications will be collected. In addition, cognitive performance, near visual acuity, anxiety as a personality trait and situational state will be evaluated.

At the end of the baseline visit, randomization to one of the two study groups will be performed. On the day of the surgical intervention, the degree of anxiety will be objectively and subjectively assessed 30 and 10 minutes before the operation for all patients. Participants in the intervention group will be shown the images 25 minutes before the operation, after the first vital signs are taken, saliva sample is collected, and the previously described scales are applied.

9. Statistical analysis: The normality of the variables will be assessed using the Kolmogorov-Smirnov test. Continuous variables will be expressed as mean ± standard deviation and qualitative variables will be expressed as number and percentage. The chi-square test will be used to analyze the association between independent qualitative variables, and the McNemar test will be used for paired samples. Comparison of means between two groups will be carried out using Student's t-test or the non-parametric Mann-Whitney U test. Change within the same group will be evaluated using a Student's t-test or the Wilcoxon test. The relationship between quantitative variables will be analyzed using the Pearson coefficient or the Spearman correlation coefficient, as appropriate. Multivariate analysis will be performed using different multiple logistic regression models to analyze the effect of the intervention. In all cases, variables that may influence the outcome, such as sociodemographic variables, drug use, presence of comorbidities, etc., will be adjusted. A bilateral hypothesis test with a risk alpha of 0.05 will be set as the limit of statistical significance. SPSS, v.25.0 will be used for the statistical analysis of the data.

10. Ethical Issues: After obtaining authorization from the Clinical Research Ethics Committee of the Salamanca health area and having previously informed the study participants, the study will be carried out in compliance with the principles of the Helsinki Declaration. Information about the project's objectives, as well as the expected benefits and risks, will be made known to the participants, and all of this will be reflected in the informed consent. Participants' confidentiality will be guaranteed at all times in accordance with the Organic Law on the Protection of Personal Data and Guarantee of Digital Rights, LO 3/2018 of December 5, and under the conditions established by the Law on Biomedical Research 14/2007.

11. Gender Perspective: In our study, the inclusion of women in the research team has been taken into account, with women making up 60% of the team. Similarly, women over the age of 18 who meet the requirements to participate in the study and voluntarily accept to participate are included in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes over 18 years of age with upper limb pathology that will be surgically treated at the University hospital complex in Salamanca.
* Signed informed consent.

Exclusion Criteria:

* Pathology to be surgically treated with a location other than the upper limb.
* Patients with a score of less than 26 points on the Mini Mental Examination (MMSE).
* Blind or visually impaired individuals who cannot correct their vision with appropriate lenses.
* Any other circumstance at the discretion of the investigators

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety level (STAI) | 1 year
  The anxiety level in both groups of patients will be measured and assessed. the validated Spanish version of Trait Anxiety Inventory will be used as an anxiety measurement scale (STAI). The scale consists of 40 items, 20 measure anxiety-trait and the other 20 anxiety-state. The minimum score is 0 points (no anxiety) and the maximum is 60 (maximum level of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: M. Pérez Saavedra, Principal Investigator — GERENCIA REGIONAL DE SALUD CASTILLA Y LEÓN

IPD SHARING:
Plan to Share IPD: No